CLINICAL TRIAL: NCT00075751
Title: A Phase II Trial of Gemcitabine, Carboplatin and PS-341 (NSC-681239) in the First-Line Treatment of Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Gemcitabine, Carboplatin, and Bortezomib in Advanced or Recurrent Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03183; S0339; U10CA032102 (NIH); CDR0000349336 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-01-09; First posted 2004-01-13 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Carboplatin; Bortezomib

ARMS (1):
- Treatment (gemcitabine hydrochloride, carboplatin, bortezomib) (Experimental): Patients receive gemcitabine IV over 30 minutes on days 1 and 8, carboplatin IV over 15-30 minutes on day 1, and bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease may continue to receive bortezomib alone on the above schedule for up to 1 year at the discretion of the treating physician.
  Interventions: Drug: gemcitabine hydrochloride; Drug: carboplatin; Drug: bortezomib

INTERVENTIONS:
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE

SUMMARY:
Phase II trial to study the effectiveness of combining bortezomib with gemcitabine and carboplatin in treating patients who have advanced or recurrent non-small cell lung cancer that has not been previously treated with chemotherapy. Drugs used in chemotherapy, such as gemcitabine and carboplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Bortezomib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Bortezomib may also help gemcitabine and carboplatin kill more tumor cells by making the cells more sensitive to the drugs

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess overall survival in chemo-naϊve patients with advanced non-small cell lung cancer (NSCLC) treated with combination of gemcitabine, carboplatin and PS-341.

SECONDARY OBJECTIVES:

I. To assess response rate (confirmed plus unconfirmed, complete plus partial), in the subset of patients with measurable disease, progression-free survival and quantitative toxicities in this group of patients treated with this regimen.

II. To investigate in an exploratory manner, the association of levels of hypoxia-induced secreted proteins and tumor DNA in plasma levels of apoptosis-associated proteins in tumor tissue, and the changes in the levels of PS-341 modulated proteins in peripheral white blood cells with patient response and survival.

OUTLINE: This is a multicenter study.

Patients receive gemcitabine IV over 30 minutes on days 1 and 8, carboplatin IV over 15-30 minutes on day 1, and bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease may continue to receive bortezomib alone on the above schedule for up to 1 year at the discretion of the treating physician.

Patients are followed every 6 months for up to 3 years after registration.

PROJECTED ACCRUAL: A total of 99 patients will be accrued for this study within 5 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically proven selected stage IIIB (T4 lesion due to malignant pleural effusion) or stage IV, advanced non-small cell lung cancer or recurrent disease after previous surgery and/or radiation
* Patients with known brain metastases are not eligible for this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events; all patients must have a pretreatment CT or MRI scan of the brain to evaluate for CNS disease within 28 days prior to registration
* Patients must have measurable OR non-measurable disease documented by CT, MRI, or x-ray; measurable disease must be assessed within 28 days prior to registration and non-measurable disease must be assessed within 42 days prior to registration; pleural effusions, ascites and laboratory parameters are not acceptable as the only evidence of disease
* Patients must not have received any prior systemic chemotherapy or biological agent for non-small cell lung cancer; prior radiation is permitted; however, two weeks must have elapsed since the completion of prior radiation therapy and patients must have recovered from all associated toxicities at the time of registration; measurable or non-measurable disease must be outside the previous radiation field or a new lesion inside the port must be present
* At least two weeks must have elapsed since surgery (thoracic or other major surgeries) and patients must have recovered from all associated toxicities at the time of registration
* Serum creatinine =< the institutional upper limit of normal OR a creatinine clearance >= 60 cc/min; these tests must have been performed within 28 days prior to registration
* ANC >= 1500/ul obtained within 14 days prior to registration
* Platelet count >= 100,000/ul obtained within 14 days prior to registration
* Serum bilirubin =< institutional upper limit of normal obtained within 28 days prior to registration
* SGOT or SGPT =< 2.5 x the institutional upper limit of normal obtained within 28 days prior to registration
* All patients must have a Zubrod performance status of 0-1
* Peripheral neuropathy, if present, must be =< grade 1 (NCI Common Terminology Criteria for Adverse Events version 3.0)
* Correlative science studies: Institutions must have IRB approval of S9925 (the Lung Cancer Specimen Repository); patients must be offered participation in S9925; with the patient's consent, tumor tissue, blood and plasma will be submitted for testing via S9925; patients must be registered separately to S9925 in order for institutions to receive credit for specimen submissions
* Patients known to be HIV positive and receiving anti-retroviral therapy (HAART) are not eligible for this study because of possible pharmacokinetic interactions
* Patients must not be planning to receive any other concomitant anticancer treatment including chemotherapy, radiation therapy, biologic agents or any other investigational drugs
* Patients should not have known hypersensitivity to boron, mannitol, or PS-341; if day 28 or 42 falls on a weekend or holiday, the limit may be extended to the next working day; in calculating days of tests and measurements, the day a test or measurement is done is considered day 0; therefore, if a test is done on a Monday, the Monday four weeks later would be considered day 28; this allows for efficient patient scheduling without exceeding the guidelines
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission or other cancer from which the patient has been disease-free for 5 years
* Pregnant or nursing women may not participate in this trial because of the increased risk of fetal harm including fetal death from the chemotherapeutic agents; women/men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* At the time of patient registration, the treating institution's name and ID number must be provided to the Data Operations Center in Seattle in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered into the data base

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2004-01; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to 3 years

SECONDARY OUTCOMES:
Response rate (confirmed plus unconfirmed, complete plus partial) | Up to 12 weeks
Progression-free survival | Up to 3 years
Toxicities, based on the National Cancer Institute Common Toxicity Criteria (NCI CTC) v3.0 | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Angela Davies, Principal Investigator — SWOG Cancer Research Network
Locations (1):
- Southwest Oncology Group, San Antonio, Texas, United States